CLINICAL TRIAL: NCT05474599
Title: Effects Of Dry Cupping Therapy on Pain and Symptoms Severity in Primary Dysmenorrhea
Brief Title: Dry Cupping Therapy And Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0522
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Primary Dysmenorrhea
Keywords: Cupping Therapies; Pain; Painful Mensturation; TENS
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry cupping therapy (Experimental): For pain and severity of symptoms in primary dysmenorrhea.
  Interventions: Other: conventional physical therapy
- Conventional physical therapy (Other): For management of pain and severity of symptoms
  Interventions: Other: Dry cupping therapy

INTERVENTIONS:
Other: conventional physical therapy — TENS
  Arms: Dry cupping therapy
Other: Dry cupping therapy — Experimental group was given Dry cupping therapy along with TENS.
  Arms: Conventional physical therapy

SUMMARY:
There is growing evidence of the effects of dry cupping therapy on pain in primary dysmenorrhea. However, very few studies have explored the effects of dry cupping therapy on the severity of symptoms in primary dysmenorrhea. The study aims to explore the effects of dry cupping therapy and the severity of symptoms in primary dysmenorrhea

DETAILED DESCRIPTION:
A randomized, standard controlled clinical trial was conducted from August 2014 to February 2016. Diagnosed case of primary dysmenorrhea aged between 12-30 years were included in the research. A total of 60 subjects were assigned randomly to the interventions. They divide subjects into three groups randomly using computer software (graph pad software quickcals) each group has 20 number of subjects .The test group A received 3gm of herbal drug namely hulba twice in a day from day 1 to day 3 of menstrual cycle. The test group B received same dose of hulba with dry cupping. For dry cupping three medium cups were applied below the umbilicus for 15 minutes on day 1 and day 3 of menstruation. Group C is controlled group which received standard drug mefanamic acid, 500 mg twice daily for same duration as the test drug. These interventions were given for three consecutive cycles by the end of three months results were analyzed. The parameters were evaluated before and after the trial. after the completion of statistical analysis they find out that the dry cupping was more effective than mefanamic acid in reducing pain intensity in dysmenorrhea .they also notice the overall improvement in other associated symptoms like nausea vomiting fatigue and headache .No adverse effects had observed either in the subjects of test group or standard group .

Another research in 2018 was conducted they divide subjects into two groups In the intervention group, dry cupping therapy from 3 days before to 3 days after the onset of menstruation for three successive menstrual cycles they placed two cups on the lower back on each side of the spine and another on the supra pubic area for 10-15 min once daily. Students in the control group did not receive cupping therapy but their PD severity symptoms were assessed and documented for three menstrual cycle .Results indicated a significant decrease in PD severity after dry cupping for three menstrual cycles. Similarly, a study in India found that cupping therapy significantly reduced the PD by improving the local blood to uterus and reduces blood congestion. This study concludes that dry cupping can be effective in significantly reducing PD and its associated symptoms. Given its effectiveness, inexpensiveness, and safety, individuals with PD can refer to cupping technicians to receive dry cupping for PD management. More studies with larger samples are still needed to provide conclusive evidence about the effectiveness of dry cupping in reducing PD .

According to research in 2018 conducted the highest incidence of PD (57.5%) was observed in the group of 15-25years and less (8.57%) in the age group of above 35 years The highest incidence of dysmenorrhea (27.5%)was observed in10th class students while lowest incidence(5%) was observed in post-graduation students. It has been concluded that cupping is very effective for relief of it is cheaper and well tolerated by patient and there are no observed side effects of cupping therapy on patient .

Reviewing the previous literature on the effects of dry cupping therapy provides sufficient evidences on pain management with Primary dysmenorrhea but controlling the other associated symptoms through dry cupping is not enough. Hence dry cupping is an effective intervention to control symptoms associated with dysmenorrhea but its clinical application is very limited. In this study dry cupping will be used to minimize pain and manage backache during menstruation.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycle
* Nulliparous

Exclusion Criteria:

* Allergic to cupping therapy,
* Endometriosis,
* PCOS
* Skin disorders

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Verbal multi-dimensional dysmenorrhea severity scoring system | 8th week
  Changes from the baseline verbal multidimensional scoring system were used. This scoring system measures pain severity and takes into account the impacts of pains on daily activities, systemic symptoms, and analgesic requirements
Numeric pain rating scale | 8th week
  Changes from baseline the Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Working Ability, Location, Intensity, Days Of Pain, Dysmenorrhea (WaLIDD) scale | 8th week
  Changes from the baseline this scale-type survey (working ability, location, intensity, days of pain, dysmenorrhea [WaLIDD] score) was designed, which integrated features of dysmenorrhea such as: 1) number of anatomical pain locations (no part of the body, lower abdomen, lumbar region, lower limbs, inguinal region), 2) Wong-Baker pain range (does not hurt, hurts a little, hurts a little more, hurts even more, hurts a lot, hurts a lot more),19 3) number of days of pain during menstruation (0, 1-2, 3-4, ≥5), and 4) frequency of disabling pain to perform their activities (never, almost never, almost always, always). Each tool's variable provided a specific score between 0 and 3, and the final score ranged from 0 to 12 points

CONTACTS AND LOCATIONS:
Overall Officials: Afifa Safdar, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Sialkot college of physical therapy, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inanmdar W, Sultana A, Mubeen U, Rahman K. Clinical efficacy of Trigonella foenum graecum (Fenugreek) and dry cupping therapy on intensity of pain in patients with primary dysmenorrhea. Chin J Integr Med. 2016 May 25. doi: 10.1007/s11655-016-2259-x. Online ahead of print. PMID 27225291
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Teheran AA, Pineros LG, Pulido F, Mejia Guatibonza MC. WaLIDD score, a new tool to diagnose dysmenorrhea and predict medical leave in university students. Int J Womens Health. 2018 Jan 17;10:35-45. doi: 10.2147/IJWH.S143510. eCollection 2018. PMID 29398923